CLINICAL TRIAL: NCT05003323
Title: Brain Biomarker of Endogenous Analgesia in Patients With Chronic Knee Pain
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Benedict Alter, Assistant Professor, University of Pittsburgh
Other Study IDs: STUDY20060254
Record Dates: First submitted 2021-08-06; First posted 2021-08-12 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Chronic Pain; Chronic Knee Pain; Knee Osteoarthritis; Analgesia
MeSH Terms: conditions — Chronic Pain; Osteoarthritis, Knee; Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High Knee Pain with Osteoarthritis: Adults 45-80 years old who have moderately severe knee osteoarthritis and rate their daily knee pain at >=6 on a 0-10 numeric rating scale
- Low Knee Pain with Osteoarthritis: Adults 45-80 who have moderately severe knee osteoarthritis and rate their daily knee pain at <=5 on a 0-10 numeric rating scale
- Healthy Controls: Age matched, BMI matched adults who do not have knee osteoarthritis or chronic pain

SUMMARY:
This case-control study in patients with knee osteoarthritis and pain-free control individuals aims to develop a brain biomarker of endogenous analgesia that may be used in subsequent clinical trials. Deficits in central nervous system (CNS) pain inhibition may contribute to chronic pain intensity, but quantitative sensory testing (QST) methods are limited. Incorporating brain imaging to assessments of CNS pain inhibition, by examining activity in relevant brain networks, would allow for an objective, physiologic measure of CNS pain inhibition. Preliminary data in pain-free volunteers implicate cortical activity measured with functional near-infrared spectroscopy (fNIRS) during CNS pain inhibition. Broadly, the investigators hypothesize that variability in CNS pain inhibition contributes to variability in clinical pain intensity.

DETAILED DESCRIPTION:
The objective of this study is to identify the neural correlates of central nervous system (CNS) pain inhibition in patients with knee osteoarthritis (OA) and determine how the correlates relate to clinical chronic (i.e., greater than 6 months) knee pain. To attain this objective, the investigators will test the following working hypotheses: (H1) in knee OA patients with moderate osteoarthritis but severe knee pain, cortical correlates of CNS pain inhibition are diminished compared to patients with less knee pain and (H2) provocation of clinical knee pain with ambulation produces greater pain-related cortical activation in patients with greater clinical knee pain at baseline. The study will also compare patients with knee OA to a control group to test the hypothesis (H3) that CNS pain inhibition behavioral and functional near-infrared spectroscopy (fNIRS) brain imaging measures are diminished in knee OA. Finally, in exploratory analysis, the investigators hypothesize that cortical functional connectivity is altered in patients with greater knee pain.

The study approach is to measure brain activity in patients with knee osteoarthritis, divided into high pain intensity and low pain intensity groups, and in pain-free controls with fNIRS scanning during rest, quantitative sensory testing (QST) measures of CNS pain inhibition (conditioned pain modulation and offset analgesia), and walking and stair climbing tasks. The rationale is that successful completion of this study will determine whether fNIRS measures relate to QST measures of CNS pain inhibition and clinical pain intensity both at rest and during activity. This fundamental knowledge, in combination with prior studies of conditioned pain modulation (CPM), will be important to understanding how CNS pain inhibition may contribute to a range of chronic pain syndromes.

ELIGIBILITY:
Inclusion Criteria:

1. For the knee arthritis groups: Chronic knee pain with evidence of knee osteoarthritis - radiographically grades 2-4
2. Age: 45-80 years old
3. Gender: Males and females will be recruited.
4. Language: only English-speaking subjects will be included.

Exclusion Criteria:

1. Inflammatory arthritis (e.g. rheumatoid arthritis)
2. Inability to walk and climb stairs unassisted
3. History of knee replacement or open knee surgery
4. History of arthroscopic knee surgery within the last 3 months (>3 months does not exclude participant)
5. History of knee radiofrequency nerve ablation or ligation
6. Current opioid use
7. Current use of antidepressants that are not in the serotonin-selective reuptake inhibitor (SSRI) class. Patients who are currently using an SSRI are allowed to take part in the study
8. Cognitive impairment affecting the ability to provide informed consent, understand directions, and participate in study procedures
9. Uncontrolled or unstable medical disorder preventing participation in study procedures
10. History of brain surgery
11. Tattoos on forearm or knee
12. Pregnancy
13. Patients with chronic pain conditions that are more severe than their knee arthritis pain (e.g., CRPS, fibromyalgia)
14. Patients whose most painful knee is excluded for another reason (e.g., recent surgery on most painful knee)
15. For the pain-free control group: a history of chronic pain
16. History of intra-articular steroid injections, platelet enriched or hyaluronic acid injections in the last 1 month

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Pitt+Me registry which comprises of any members of the local population who are registered in the program.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Differences in offset analgesia | 15 minutes
  Pain intensity difference during offset and control heat stimuli
Differences in brain region activation- QST | 2-3 hours
  Difference in brain region activation (as measured by oxygenated hemoglobin, HbO) between CNS inhibition and control stimuli during QST procedures.
Differences in brain region activation- walking test | 15 minutes
  Change in brain region activation (HbO) between rest and ambulation during the 6 minute walking test test
Differences in brain region activation- stair climbing | 15 minutes
  Change in brain region activation (HbO) between rest and ambulation during the stair climbing test

SECONDARY OUTCOMES:
Differences in resting fNIRS signaling | 5-10 minutes
  Differences in fNIRS resting state connectivity as measured by brain region activation
QST battery responses | 2-3 hours
  Differences in responses to QST to characterize threshold and tolerance to cutaneous thermal and mechanical stimuli
Pain intensity scores after stair climbing task | 10 minutes
  Verbal score from 0-100 on numeric rating scale (NRS) of pain following stair climbing task. Higher NRS scores indicate higher pain intensity.
Pain intensity scores after walking test | 6 minutes
  Verbal score from 0-100 on NRS of pain following 6 minute walking task. Higher NRS scores indicate higher pain intensity.
Duration of stair climbing task | 10 minutes
  Differences in time taken to complete stair climbing task
Distance walked during 6 minute walking task | 6 minutes
  Differences in distance walked during 6 minute walking task
Questionnaire score- PROMIS 29 | 1 hour
  Standardized survey score of PROMIS-29 assessing physical and mental health. Physical Function Score ranges from 4-20. Anxiety Score ranges from 4-20. Depression Score ranges from 4-20. Fatigue Score ranges from 4-20. Sleep Disturbance Score ranges from 4-20. Social Roles Score ranges from 4-20. Pain Interference Score ranges from 4-20. Pain Intensity Score ranges from 0-10. Higher scores indicate worse mental and physical health.
Questionnaire score- Knee Injury and Osteoarthritis Outcome Score (KOOS) | 1 hour
  Standardized survey called Knee Injury and Osteoarthritis Outcome Score assessing knee pain. Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.
Questionnaire score- State Trait Anxiety Inventory (STAI) Y1-2 | 1 hour
  Standardized survey score of state trait anxiety inventory Y1 and Y2 assessing anxiety before QST procedures.
  State Anxiety Score ranges from 20-80. Trait Anxiety Score ranges from 20-80. Higher scores indicate worse anxiety state and trait symptoms.
Questionnaire score- Pain Catastrophizing Scale (PCS) | 1 hour
  Standardized survey score assessing pain perception before QST procedures. Rumination subscale score ranges from 0-16. Magnification subscale score ranges 0-12. Helplessness subscale score ranges from 0-24. Total score can be calculated by summing subscales. Total score ranges from 0-52, with higher scores indicating more pain catastrophizing.
Questionnaire score- STAI Y1 post testing | 1 hour
  Standardized survey score of state trait anxiety inventory Y1 assessing anxiety immediately after QST procedures. Higher scores indicate worse anxiety state.
Questionnaire score- Situational Pain Catastrophizing Scale post testing | 1 hour
  Standardized survey score assessing pain perception immediately after QST procedures are completed.
  Scores range from 0-24, with higher scores representing more pain catastrophizing.
Questionnaire score- Situational Pain Catastrophizing Scale post mobility tasks | 1 hour
  Standardized survey score assessing pain perception immediately after walking and stair climbing tasks are completed.
  Scores range from 0-24, with higher scores representing more pain catastrophizing.
Questionnaire score- Beck Depression Inventory-II (BDI-II) | 1 hour
  Standardized survey assessing depression. Scores range from 0-63. Total score of 0-13 is considered minimal range of depression, 14-19 is mild, 20-28 is moderate, and 29-63 is severe depression.
Questionnaire score- Generalized Anxiety Disorder 2-item (GAD-2) | 1 hour
  Standardized survey score of GAD-2 assessing anxiety. Scores range from 0-6. Higher scores indicate higher likelihood of having GAD.
Questionnaire score- Barratt Impulsiveness Scale-11 | 1 hour
  Standardized survey score of Barratt Impulsiveness Scale-11 assessing the personality/behavioral construct of impulsiveness.
  Attention Impulsiveness Score ranges from 8-32. Motor Impulsiveness Score ranges from 11-44. Non-planning Impulsiveness Score ranges from 11-44. Subscale scores can be summed for a total score. Higher scores indicate greater levels of impulsivity.
Questionnaire score- Barratt Simplified Measure of Social Status | 1 hour
  Standardized survey score of Barratt Simplified Measure of Social Status that measures social status based on marital status, employment status, educational attainment, and occupational prestige. Total Education Score ranges from 3-21. Total Occupation Score ranges from 5-45. Total score of education and occupation can be calculated by summing the subscales with a range 8-66. Higher scores indicate a higher social status.
Questionnaire score- Patient Health Questionnaire 2 (PHQ-2) | 1 hour
  The PHQ-2 inquires about the frequency of depressed mood and anhedonia over the past two weeks. The PHQ-2 includes the first two items of the PHQ-9. A PHQ-2 score ranges from 0-6. The authors identified a score of 3 as the optimal cutpoint when using the PHQ-2 to screen for depression.
  If the score is 3 or greater, major depressive disorder is likely.
Questionnaire score- Fibromyalgia Severity Scale | 1 hour
  This questionnaire tests if patients meet the 2016 criteria for fibromyalgia. The symptom severity score ranges from 0-12, with higher scores indicating a higher likelihood of fibromyalgia. Three symptom question items range from 0-3, and these are summed up for the final score (totaling 0-9). Three additional symptom questions have yes or no options. If the patient answers yes, 1 point is added to the final scale.

CONTACTS AND LOCATIONS:
Overall Officials: Benedict Alter, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Pain Medicine at Centre Commons, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alter BJ, Maurer M, O'Connell B, Sanchez AG, Kaynar AM, DiGioia AM, Huppert T, Wasan AD. Deficits in temporal pain inhibition are associated with greater pain and functional impairment in osteoarthritis. Pain. 2025 Nov 1;166(11):2490-2509. doi: 10.1097/j.pain.0000000000003648. Epub 2025 Jun 19. PMID 40539481